CLINICAL TRIAL: NCT04051086
Title: Quantification of Elastin Markers Synthesis in Williams-Beuren Syndrome and 7q11.23 Micro-duplication Syndrome
Acronym: ELAST7
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0368
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Williams-Beuren Syndrome; Micro-duplication 7q11.23 Syndrome; Vasculopathy
Keywords: Williams-Beuren Syndrome; Micro-duplication 7q11.23 syndrome; Vasculopathy
MeSH Terms: conditions — Williams Syndrome; Vascular Diseases | interventions — Restraint, Physical; Urination; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Williams Beuren (Other): Subjects aged from 3 months to 60 years with a diagnosis confirmed with FISH of Williams Beuren syndrome.
  Interventions: Biological: Physical examination and Urine and blood samples
- Micro-duplication 7q11.23 (Other): Subjects aged from 3 months to 60 years with a diagnosis confirmed with CGHarray of micro-duplication 7q11.23 syndrome.
  Interventions: Biological: Physical examination and Urine and blood samples
- Healthy Group (Other): Subjects without cardiovascular and neurological medical history.
  Interventions: Biological: Urine and blood samples

INTERVENTIONS:
Biological: Physical examination and Urine and blood samples — Only one visit for each participant : A large majority of visits will be part of patients' usual care
  * Medical examination : birth, weight, gender, blood pressure, medical history
  * Urine and blood samples
  Arms: Micro-duplication 7q11.23; Williams Beuren
Biological: Urine and blood samples — Only one visit for each participant
  * Medical history
  * Urine and blood samples
  Arms: Healthy Group

SUMMARY:
Introduction: Williams-Beuren syndrome is a rare genetic disorder caused by a 7q11.23 microdeletion. The phenotype associates vasculopathy (arterial stenosis, hypertension), dimorphism and intellectual disability. Microdeletion includes several genes: ELN encodes for elastin and the haplo-insufficiency (only 1 functional copy) causes vasculopathy.

The primary objective is to quantify plasma and urinary levels of elastin peptides in Williams-Beuren patients and 7q11.23 micro-duplication syndrome patients in order to correlate the levels of these markers with the number of copies of ELN gene (proportional positive relationship "gene copy number - circulating levels of markers) Materials and Methods: This prospective study will be carried out in Lyon at the "Hôpital Femme-Mère-Enfant" for 2 years. 3 groups of patients will be studied: Williams-Beuren patients (N=20), micro-duplication 7q11.23 syndrome patients (N=10) and healthy patients (N=60). Subjects will be followed for 1 day.

Clinical examination (weight, height, blood pressure) and biological sample collection (blood and urine sample) will be carry out for Williams Beuren and micro-duplication 7q11.23 patients group. A large majority of visits will be part of patients' usual care. A large part of patients are systematically seen in consultation once a year. For healthy group, only biological sample collection will be carry out. The PE concentrations will be assessed and compared between the three groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age : from 3 months to 60 years old
* Williams Beuren group : Diagnosis confirmed with FISH
* Micro-duplication 7q11.23 group : Diagnosis confirmed with CGHarray
* Healthy Group : no cardiovascular and neurological medical history
* Informed consent

Exclusion Criteria:

* No social insurance
* Subject under judicial protection
* Subject participating in another research including an exclusion period still in progress

Ages: 3 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Plasma level of elastin peptides (PE) | 1 day
  To quantify plasma level of elastin peptides in participants in order to correlate the levels of these markers with the number of copies of ELN gene (proportional positive relationship "gene copy number - circulating levels of markers).
  The primary endpoint will be assessed by measuring the blood level of PE between groups
Urinary level of elastin peptides (PE) | 1 day
  To quantify urinary level of elastin peptides in participants in order to correlate the levels of these markers with the number of copies of ELN gene (proportional positive relationship "gene copy number - circulating levels of markers).
  The primary endpoint will be assessed by measuring the urinary level of PE between groups

SECONDARY OUTCOMES:
Correlation between blood level of PE and cardiovascular involvement in patients. | 1 day
  Blood level of PE will be correlated with the presence / severity of cardiovascular disease
Correlation between urinary level of PE and cardiovascular involvement in patients. | 1 day
  Urinary level of PE will be correlated with the presence / severity of cardiovascular disease
Blood level of PE in treated and untreated minoxidil patients | 1 day
  Blood levels of PE in the samples of patients who participated in the minoxidil clinical trial will be compare to those of participants of this study
Urinary level of PE in treated and untreated minoxidil patients | 1 day
  Urinary levels of PE in the samples of patients who participated in the minoxidil clinical trial will be compare to those of participants of this study

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No